CLINICAL TRIAL: NCT04391322
Title: Assessment of CFTR-Modulator Treatment in Cystic Fibrosis Lung Disease Using Novel Structural and Functional MRI
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000063021
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Group 1: Healthy Controls; Group 2: Stable CF; Group 3: CF Participants Anticipated to Receive CFTR-modulator Therapy; Group 4: 4-8 yo CF Participants Starting Triple Combination Modulator Therapy
Keywords: CFTR modulator treatment; xenon MRI; Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Healthy participants without lung disease
- Group 2: Participants with stable cystic fibrosis
- Group 3: Participants with cystic fibrosis, anticipated to receive treatment with CFTR-modulator therapy. Please note: treatment is determined by your physician as part of your normal therapy plan.
- Group 4: Participants with CF who are between 4-8 years old and are starting triple combination modulator therapy using the rapid lung and abdominal imaging methods.

SUMMARY:
This is a prospective, longitudinal observational study conducted at The Hospital for Sick Children (SickKids). The purpose of this study is to evaluate the ability of MRI to detect changes in lung structure and function in CF patients receiving CFTR-modulator therapy. Participants who meet eligibility criteria and consent to the study will undergo study procedures which include spirometry and body plethysmography (optional), multiple breath washout testing, MRI and measurement of quality of life. The study will consist of three to six study visits for Group 1, 2 and 3: baseline, one month (±1 week) and 6 month (±2 week) and if they re-consent then 3 additional visits of 1 year (±6 months). (2 years (±6 months) and 3 years (±6 months) follow-up. Some participants in Group 2 may transition to Group 3.

This study includes three populations of interest: Group 1: 25 healthy volunteers, Group 2: 25 patients with stable CF lung disease , Group 3: 20 patients with CF lung disease anticipated to receive treatment with CFTR-modulator therapy and Group 4: 18 patients with CF who are between 4-8 years old and are starting triple combination modulator therapy using the rapid lung and abdominal imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to 4 years of age
* Informed consent by patient or parent/guardian consent and participant assent when appropriate.
* Able to perform reproducible spirometry and achieve a breath hold duration sufficient for MRI acquisition

Exclusion Criteria:

* Medical instability that would preclude the ability to undergo the required investigations
* FEV1 % predicted < 40%
* Severe claustrophobia
* Does not meet MRI screening criteria
* Cough within the past 3 days prior to study visit
* Usage of oral antibiotics within 3 weeks prior to study visit

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study includes four populations of interest: Group 1: 25 healthy volunteers, Group 2: 25 patients with stable CF lung disease and Group 3: 20 patients with CF lung disease anticipated to receive treatment with CFTR-modulator therapy and Group 4: 18 patients with CF who are between 4-8 years old and are starting triple combination modulator therapy using the rapid lung and abdominal imaging methods
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reproducibility | 36 months
  Establish the interscan reproducibility of fractional ventilation maps and 1H MRI over three and up to six visits in healthy volunteers and in patients with stable CF lung disease and compare to conventional spirometry and LCI.
Correlation | 12 months
  Correlate changes in lung structure and function detected by MRI imaging with clinical outcomes including FEV1 rate of decline, frequency of pulmonary exacerbations, days of IV antibiotics and hospital days to treat pulmonary exacerbation and change in health-related quality of life measures (CFQ-R scores and CF-QUEST) in the setting of patients with stable CF lung disease and those receiving CFTR-modulator therapy.
Responsiveness | 36 months
  Assess responsiveness of MRI to treatment effects over three and up to six visits visits in CF patients receiving CFTR-modulator therapy and compare to conventional breathing tests
Younger cohort | 24 months
  Extension of above objectives originally only explored in children ages 8-18 years old, to younger cohort of CF participants ages 4-8 years old at baseline prior to initiation of CFTR modulator therapy, as well as at 12 and 24 months after therapy initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared between the two participating sites in the study. A data transfer agreement has been implemented to enable this transfer smoothly.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after enrolling the first participant and will be available for the duration of the study